CLINICAL TRIAL: NCT01703000
Title: NG PROMUS: A Prospective, Multicenter Trial to Assess the NG PROMUS Everolimus-Eluting Platinum Chromium Coronary Stent System (NG PROMUS Stent System) for the Treatment of Atherosclerotic Lesion(s)
Brief Title: NG PROMUS Stent System for the Treatment of Atherosclerotic Coronary Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NG PROMUS Clinical Trial S2294
Record Dates: First submitted 2012-10-05; First posted 2012-10-10 (Estimated); Results first posted 2014-03-21 (Estimated); Last update posted 2014-04-15 (Estimated); Status verified 2014-03

CONDITIONS: Atherosclerosis; Coronary Artery Disease
Keywords: drug eluting coronary stent
MeSH Terms: conditions — Atherosclerosis; Coronary Artery Disease | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NG PROMUS stent (Experimental): Single-arm treatment group receiving interventional NG PROMUS study stent
  Interventions: Device: Percutaneous coronary intervention (NG PROMUS)

INTERVENTIONS:
Device: Percutaneous coronary intervention (NG PROMUS) — Interventional coronary artery stenting with NG PROMUS study stent.

SUMMARY:
NG PROMUS: A Prospective, Multicenter Trial to Assess the NG PROMUS Everolimus-Eluting Platinum Chromium Coronary Stent System (NG PROMUS Stent System) for the Treatment of Atherosclerotic Lesion(s)

DETAILED DESCRIPTION:
To evaluate clinical and peri-procedural angiographic and intravascular ultrasound (IVUS) outcomes for the NG PROMUS Everolimus-Eluting Platinum Chromium Coronary Stent System (NG PROMUS Stent System) in the treatment of subjects with atherosclerotic lesion(s) ≤ 34 mm in length (by visual estimate) in native coronary arteries ≥ 2.50 mm to ≤ 4.0 mm in diameter (by visual estimate)

ELIGIBILITY:
Clinical Inclusion Criteria:

1. Subject must be at least 18 years of age
2. Subject (or legal guardian) understands the trial requirements and the treatment procedures and provides written informed consent before any trial-specific tests or procedures are performed
3. Subject is eligible for percutaneous coronary intervention (PCI)
4. Subject has symptomatic coronary artery disease with objective evidence of ischemia or silent ischemia
5. Subject is an acceptable candidate for coronary artery bypass grafting (CABG)
6. Subject is willing to comply with all protocol-required follow-up evaluation

Angiographic Inclusion Criteria:

1. Target lesion(s) must be located in a native coronary artery with a visually estimated reference vessel diameter (RVD) ≥2.50 mm and ≤4.0 mm
2. Target lesion(s) length must be ≤34 mm (by visual estimate)
3. Target lesion(s) must have visually estimated stenosis ≥50% and <100% with thrombolysis in Myocardial Infarction (TIMI) flow >1 and one of the following (stenosis ≥70%, abnormal fractional flow reserve (FFR), abnormal stress test or imaging stress test, or elevated biomarkers) prior to procedure
4. Coronary anatomy is likely to allow delivery of a study device to the target lesions(s)
5. The first lesion treated must be successfully pre-dilated/pretreated Note: Successful pre-dilatation/pretreatment refers to dilatation with a balloon catheter of appropriate length and diameter, or pretreatment with directional or rotational coronary atherectomy, laser or cutting/scoring balloon with no greater than 50% residual stenosis and no dissection greater than National Heart, Lung, Blood Institute (NHLBI) type C.

Clinical Exclusion Criteria:

1. Subject has clinical symptoms and/or electrocardiogram (ECG) changes consistent with acute ST elevation MI (STEMI)
2. Subject has cardiogenic shock, hemodynamic instability requiring inotropic or mechanical circulatory support, intractable ventricular arrhythmias, or ongoing intractable angina
3. Subject has received an organ transplant or is on a waiting list for an organ transplant
4. Subject is receiving or scheduled to receive chemotherapy within 30 days before or after the index procedure
5. Planned PCI (including staged procedures) or CABG after the index procedure
6. Subject previously treated at any time with intravascular brachytherapy
7. Subject has a known allergy to contrast (that cannot be adequately premedicated) and/or the trial stent system or protocol-required concomitant medications (e.g., platinum, platinum-chromium alloy, stainless steel, everolimus or structurally related compounds, polymer or individual components, all P2Y12 inhibitors, or aspirin)
8. Subject has one of the following (as assessed prior to the index procedure):Other serious medical illness (e.g., cancer, congestive heart failure) with estimated life expectancy of less than 24 months; Current problems with substance abuse (e.g., alcohol, cocaine, heroin, etc.);Planned procedure that may cause non-compliance with the protocol or confound data interpretation
9. Subject is receiving chronic (≥72 hours) anticoagulation therapy (i.e., heparin, coumadin) for indications other than acute coronary syndrome
10. Subject has a platelet count <100,000 cells/mm3 or >700,000 cells/mm3
11. Subject has a white blood cell (WBC) count < 3,000 cells/mm3
12. Subject has documented or suspected liver disease, including laboratory evidence of hepatitis
13. Subject is on dialysis or has baseline serum creatinine level >2.0 mg/dL (177µmol/L)
14. Subject has a history of bleeding diathesis or coagulopathy or will refuse blood transfusions
15. Subject has had a history of cerebrovascular accident (CVA) or transient ischemic attack (TIA) within the past 6 months
16. Subject has an active peptic ulcer or active gastrointestinal (GI) bleeding
17. Subject has signs or symptoms of active heart failure (i.e., NYHA class IV) at the time of the index procedure
18. Subject is participating in another investigational drug or device clinical trial that has not reached its primary endpoint
19. Subject intends to participate in another investigational drug or device clinical trial within 12 months after the index procedure
20. Subject with known intention to procreate within 12 months after the index procedure (women of child-bearing potential who are sexually active must agree to use a reliable method of contraception from the time of screening through 12 months after the index procedure)
21. Subject is a woman who is pregnant or nursing (a pregnancy test must be performed within 7 days prior to the index procedure in women of child-bearing potential)

Angiographic Exclusion Criteria:

1. Planned treatment of more than 3 lesions.
2. Planned treatment of lesions in more than 2 major epicardial vessels
3. Planned treatment of a single lesion with more than 1 stent
4. Subject has 2 target lesions in the same vessel that are separated by less than 15 mm (by visual estimate)
5. Target lesion(s) is located in the left main
6. Target lesion(s) is located within 3 mm of the origin of the left anterior descending (LAD) coronary artery or left circumflex (LCx) coronary artery by visual estimate.
7. Target lesion(s) is located within a saphenous vein graft or an arterial graft
8. Target lesion(s) will be accessed via a saphenous vein graft or arterial graft
9. Target lesion(s) with a TIMI flow 0 (total occlusion) or TIMI flow 1 prior to guide wire crossing
10. Target lesion(s) treated during the index procedure that involves a complex bifurcation (e.g., bifurcation lesion requiring treatment with more than 1 stent)
11. Target lesion(s) is restenotic from a previous stent implantation or study stent would overlap with a previous stent
12. Subject has unprotected left main coronary artery disease (>50% diameter stenosis)
13. Subject has been treated with any type of PCI (i.e., balloon angioplasty, stent, cutting balloon atherectomy) within 24 hours prior to the index procedure
14. Thrombus, or possible thrombus, present in the target vessel (by visual estimate)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-11; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John A Ormiston, MBChB, FRACP, FRACR, Principal Investigator — Mercy Angiography Unit, Ltd. Mercy Hospital
Locations (9):
- Fremantle Hospital, Fremantle, Western Australia, Australia
- New Zealand (6):
  - Mercy Angiography Unit, Ltd. Mercy Hospital, Auckland
  - Auckland City Hospital, Auckland
  - North Shore Hospital, Auckland
  - Ascot Angiography, Auckland
  - Christchurch, Christchurch
  - Middlemore Hospital, Otahuhu
- Singapore (2):
  - National University Hospital Singapore, Singapore
  - National Heart Center Singapore, Singapore

REFERENCES:
- See also: Drug-eluting product information from Manufacturer — http://www.pharma.us.novartis.com/info/products/name/zortress.jsp

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment of subjects for NG PROMUS study started on November 20, 2012 and completed on March 12, 2013. Subjects were recruited at 9 investigational centers in Australia, New Zealand and Singapore.
Period: Overall Study
Arm/Group | NG PROMUS Stent
Started | 100
Completed | 99
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Population: Single arm with investigational NG PROMUS Everolimus Eluting Coronary Stent System
  N=100 patients, N=119 Lesions, N=127 Stents
Arm/Group | NG PROMUS Stent
Number analyzed (Participants) | 100
Age, Customized [Mean (Standard Deviation); unit: years] | 61.72 (9.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 85
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 2
  Caucasian | 72
  Asian | 13
  Black, of African Heritage | 1
  Native Hawaiian or Other Pacific Islander | 5
  Other | 6
  Not disclosed | 1
Region of Enrollment [Number; unit: participants]
  Singapore | 10
  Australia | 2
  New Zealand | 88
Cardiac History [Number; unit: participants] — Note: A single participant could potentially experience multiple categories listed below.
  participants
    Previous Percutaneous Coronary Intervention | 23
    Previous Coronary Artery Bypass Graft | 5
    Previous Myocardial Infarction | 16
    Congestive Heart Failure | 2
    Stable Angina | 51
    Unstable Angina | 25
    Silent Ischemia | 7
Cardiac Risk Factors [Number; unit: participants] — Note: A single participant could potentially experience multiple categories listed below.
  participants
    Smoking, Ever | 56
    Medically Treated Diabetes | 16
    Hyperlipidemia Requiring Medication | 78
    Hypertension Requiring Medication | 70
    Family History of Coronary Artery Disease | 51
Lesion Characteristics: Target Lesion Vessel [Number; unit: Lesions] — Note: A single participant could potentially experience multiple categories listed below.
  Lesions
    Left Anterior Descending Artery | 60
    Circumflex Artery | 27
    Right Coronary Artery | 32
Lesion Characteristic: Lesion Location [Number; unit: Lesions] — Note: A single participant could potentially experience multiple categories listed below.
  Lesions
    Ostial | 8
    Proximal | 47
    Mid | 49
    Distal | 15
Lesion Characteristic: Lesion Length [Number; unit: Lesions] — Note: A single participant could potentially experience multiple categories listed below.
  Lesions
    Less than or equal to 20 mm | 91
    Greater than 20 mm | 28
Lesion Characteristics [Number; unit: Lesions] — Note: A single participant could potentially experience multiple categories listed below.
  Lesions
    Tortuosity, Any | 10
    Calcification, Any | 35
    Ulcerated | 3
    Aneurysm | 2
    Bifurcation | 61
    Total Occlusion | 2
    Eccentric Lesion | 86
Lesion Characteristic: Pre-Procedure Thrombolysis in Myocardial Infarction (TIMI) Flow [Number; unit: Lesions] — Note: A single participant could potentially experience multiple categories listed below.
  Lesions
    0 (no perfusion) | 0
    1 (penetration with minimal perfusion) | 2
    2 (partial perfusion) | 9
    3 (complete perfusion) | 108
Lesion Characteristics by Quantitative Cornary Angiography [Mean (Standard Deviation); unit: Millimeters]
  Reference Vessel Diameter | 2.78 (0.45)
  Minimum Lumen Diameter | 0.85 (0.29)
  Lesion Length | 16.05 (7.14)
Lesion Characteristic: Percent Diameter Stenosis by QCA [Mean (Standard Deviation); unit: Percent Diameter Stenosis] | 69.12 (9.69)

OUTCOME MEASURES:

1. Primary Outcome: Technical Success Rate
Description: Technical success is defined as successful delivery and deployment of the study stent to the target lesion, without balloon rupture or stent embolization, and post-procedure diameter stenosis of <30% assessed in 2 near-orthogonal projections with TIMI 3 flow in the target lesion, as visually assessed by the physician
Time Frame: Participants will be followed for the duration of hospital stay, an expected average of 1 day
Measure: Number (95% Confidence Interval); unit: percentage of lesions
Units Other Than Participants: Lesions
Arm/Group | NG PROMUS Stent
Number analyzed (Participants) | 100
Number analyzed (Lesions) | 119
percentage of lesions | 99.2 [95.4 to 100]

2. Secondary Outcome: Target Lesion Revascularization (TLR) Rate
Description: Target lesion revascularization is any ischemia-driven repeat percutaneous intervention, to improve blood flow, of the successfully treated target lesion or bypass surgery of the target vessel with a graft distally to the successfully treated target lesion. A TLR will be considered as ischemia-driven if the target lesion diameter stenosis is >/= 50% by QCA and there is presence of clinical or functional ischemia which cannot be explained by other coronary or graft lesions. Clinical or functional ischemia is any of the following:
  * The subject has a positive functional study corresponding to the area served by the target lesion.
  * The subject has ischemic ECG changes at rest in a distribution consistent with the target vessel.
  * The subject has ischemic symptoms referable to the target lesion. A TLR will be considered as ischemia-driven if the lesion diameter stenosis is >/= 70% by QCA even in the absence of clinical or functional ischemia.
Time Frame: Participants will be followed for the duration of hospital stay, an expected average of 1 day and at 30 days
Measure: Number; unit: percentage of participants
Arm/Group | NG PROMUS Stent
Number analyzed (Participants) | 100
percentage of participants | 0

3. Secondary Outcome: Target Lesion Failure (TLF) Rate
Description: Target lesion failure is any ischemia-driven revascularization of the target lesion, MI (Q-wave and non-Q-wave) related to the target vessel, or (cardiac) death. For the purposes of this protocol, if it cannot be determined with certainty whether the MI was related to the target vessel, it will be considered a TLF.
  The MI definition used for Target Lesion Failure was the PLATINUM MI definition.
Time Frame: Participants will be followed for the duration of hospital stay, an expected average of 1 day and at 30 days
Measure: Number; unit: percentage of participants
Arm/Group | NG PROMUS Stent
Number analyzed (Participants) | 100
percentage of participants | 2

4. Secondary Outcome: Target Vessel Revascularization (TVR) Rate
Description: Target vessel revascularization is defined as a TLR or a TVR remote. Target vessel revascularization remote is any ischemia-driven repeat percutaneous intervention, to improve blood flow, or bypass surgery of not previously existing lesions diameter stenosis >/= 50% by QCA in the target vessel, excluding the target lesion. A TVR will be considered ischemia-driven if the target vessel diameter stenosis is >/= 50% by QCA and any of the following are present:
  * The subject has a positive functional study corresponding to the area served by the target vessel.
  * The subject has ischemic ECG changes at rest in a distribution consistent with the target vessel.
  * The subject has ischemic symptoms referable to the target vessel. A TVR will also be considered as ischemia-driven if the lesion diameter stenosis is >/=70% even in the absence of clinical or functional ischemia.
Time Frame: Participants will be followed for the duration of hospital stay, an expected average of 1 day and at 30 days
Measure: Number; unit: percentage of participants
Arm/Group | NG PROMUS Stent
Number analyzed (Participants) | 100
percentage of participants | 0

5. Secondary Outcome: Target Vessel Failure (TVF) Rate
Description: Target vessel failure is any ischemia-driven revascularization of the target vessel, MI (Q-wave and non-Q-wave) related to the target vessel or death related to the target vessel. For the purposes of this protocol, if it cannot be determined with certainty whether the MI or death was related to the target vessel, it will be considered a TVF.
  The MI definition used was the PLATINUM MI definition.
Time Frame: Participants will be followed for the duration of hospital stay, an expected average of 1 day and at 30 days
Measure: Number; unit: percentage of participants
Arm/Group | NG PROMUS Stent
Number analyzed (Participants) | 100
percentage of participants | 2

6. Secondary Outcome: Myocardial Infarction (MI, Q-wave and Non-Q-wave) Rate
Description: MI will be defined according to the PLATINUM Definition of MI with evidence pre-specified for i) Spontaneous, ii) PCI-related, iii) CABG related, and iv) autopsy evidence criteria.
Time Frame: Participants will be followed for the duration of hospital stay, an expected average of 1 day and at 30 days
Measure: Number; unit: percentage of participants
Arm/Group | NG PROMUS Stent
Number analyzed (Participants) | 100
percentage of participants | 1

7. Secondary Outcome: Cardiac Death Rate
Description: Cardiac death is defined as death due to any of the following.
  * Acute MI
  * Cardiac perforation/pericardial tamponade
  * Arrhythmia or conduction abnormality
  * CVA through hospital discharge or CVA suspected of being related to the procedure
  * Death due to complication of the procedure, including bleeding, vascular repair, transfusion reaction, or bypass surgery
  * Any death in which a cardiac cause cannot be excluded
Time Frame: Participants will be followed for the duration of hospital stay, an expected average of 1 day and at 30 days
Measure: Number; unit: percentage of participants
Arm/Group | NG PROMUS Stent
Number analyzed (Participants) | 100
percentage of participants | 1

8. Secondary Outcome: Non-cardiac Death Rate
Description: Non-cardiac death is defined as a death not due to any of the following:
  * Acute MI
  * Cardiac perforation/pericardial tamponade
  * Arrhythmia or conduction abnormality
  * CVA through hospital discharge or CVA suspected of being related to the procedure
  * Death due to complication of the procedure, including bleeding, vascular repair, transfusion reaction, or bypass surgery
  * Any death in which a cardiac cause cannot be excluded
Time Frame: Participants will be followed for the duration of hospital stay, an expected average of 1 day and at 30 days
Measure: Number; unit: percentage of participants
Arm/Group | NG PROMUS Stent
Number analyzed (Participants) | 100
percentage of participants | 0

9. Secondary Outcome: All Death Rate
Description: Death is categorized as cardiac or non-cardiac deaths.
Time Frame: Participants will be followed for the duration of hospital stay, an expected average of 1 day and at 30 days
Measure: Number; unit: percentage of participants
Arm/Group | NG PROMUS Stent
Number analyzed (Participants) | 100
percentage of participants | 1

10. Secondary Outcome: Cardiac Death or MI Rate
Description: Any cardiac death or MI event meeting the criteria defined for a cardiac death or MI.
  MI definition used was the PLATINUM definition for MI.
Time Frame: Participants will be followed for the duration of hospital stay, an expected average of 1 day and at 30 days
Measure: Number; unit: percentage of participants
Arm/Group | NG PROMUS Stent
Number analyzed (Participants) | 100
percentage of participants | 2

11. Secondary Outcome: All Death or MI Rate
Description: Any all-cause mortality event or MI meeting the criteria defined for any death or MI.
  MI definition used was the PLATINUM definition for MI.
Time Frame: Participants will be followed for the duration of hospital stay, an expected average of 1 day and at 30 days
Measure: Number; unit: percentage of participants
Arm/Group | NG PROMUS Stent
Number analyzed (Participants) | 100
percentage of participants | 2

12. Secondary Outcome: All Death/MI/TVR Rate
Description: Any event meeting the pre-specified criteria for any death, MI, or TVR.
  MI definition used was the PLATINUM definition for MI.
Time Frame: Participants will be followed for the duration of hospital stay, an expected average of 1 day and at 30 days
Measure: Number; unit: percentage of participants
Arm/Group | NG PROMUS Stent
Number analyzed (Participants) | 100
percentage of participants | 2

13. Secondary Outcome: Stent Thrombosis Rate (by Academic Research Consortium [ARC] Definitions)
Description: Stent thrombosis should be reported as a cumulative value at the different time points and with the different separate time points. Time 0 is defined as the time point after the guide catheter has been removed and the patient left the catheterization lab.
  Timing:
  * Acute stent thrombosis*: 0 24 hours after stent implantation
  * Subacute stent thrombosis*: >24 hours to 30 days after stent implantation
  * Late stent thrombosis: >30 days to 1 year after stent implantation
  * Very late stent thrombosis: >1 year after stent implantation * Acute/subacute can also be replaced by early stent thrombosis. Early stent thrombosis is 0 30 days.
  Stent thrombosis may be defined as:
  * Confirmed/definite
  * Probable
  * Possible
  Confirmed/Definite (is considered either angiographic confirmed or pathologic confirmed)
Time Frame: Participants will be followed for the duration of hospital stay, an expected average of 1 day and at 30 days
Measure: Number; unit: percentage of participants
Arm/Group | NG PROMUS Stent
Number analyzed (Participants) | 100
percentage of participants | 0

14. Secondary Outcome: Clinical Procedural Success Rate
Description: Clinical procedural success is post-procedure diameter stenosis <30% in 2 near-orthogonal projections with TIMI 3 flow in all target lesions, as visually assessed by the physician, without the occurrence of in-hospital MI, TVR, or cardiac death.
  MI definition used was the PLATINUM definition for MI.
Time Frame: Participants will be followed for the duration of hospital stay, an expected average of 1 day
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | NG PROMUS Stent
Number analyzed (Participants) | 100
percentage of participants | 99 [94.6 to 100]

15. Secondary Outcome: In-stent Percent Diameter Stenosis (%DS)
Description: As measured by an independent angiographic core laboratory using quantitative coronary angiography (QCA), the % diameter stenosis of the in-stent region.
  Percent diameter stenosis: Relative changes that occur in the percent diameter stenosis are provided by the following relationship: % diameter stenosis= (1-[Minimum Lumen Diameter/Reference diameter]) x 100.
Time Frame: Participants will be followed for the duration of hospital stay, an expected average of 1 day
Measure: Mean (Standard Deviation); unit: In-Stent % Diameter Stenosis
Units Other Than Participants: Lesions
Arm/Group | NG PROMUS Stent
Number analyzed (Participants) | 100
Number analyzed (Lesions) | 119
In-Stent % Diameter Stenosis | 3.86 (8.43)

16. Secondary Outcome: In-segment Percent Diameter Stenosis (%DS)
Description: As measured by an independent angiographic core laboratory using quantitative coronary angiography (QCA), the % diameter stenosis of the in-segment region (in-segment includes the stented region and 5 mm edge regions).
  Percent diameter stenosis: Relative changes that occur in the percent diameter stenosis are provided by the following relationship: % diameter stenosis= (1-[Minimum Lumen Diameter/Reference diameter]) x 100.
Time Frame: Participants will be followed for the duration of hospital stay, an expected average of 1 day
Measure: Mean (Standard Deviation); unit: Diameter Stenosis, In-Segment (%)
Units Other Than Participants: Lesions
Arm/Group | NG PROMUS Stent
Number analyzed (Participants) | 100
Number analyzed (Lesions) | 119
Diameter Stenosis, In-Segment (%) | 18.14 (7.9)

17. Secondary Outcome: In-stent Minimum Lumen Diameter (MLD)
Description: As measured by an independent angiographic core laboratory using quantitative coronary angiography (QCA); the minimum lumen diameter (MLD) measured at the in-stent region.
  The MLD is the mean minimum lumen diameter (mm) from 2 orthogonal views.
Time Frame: Participants will be followed for the duration of hospital stay, an expected average of 1 day
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Lesions
Arm/Group | NG PROMUS Stent
Number analyzed (Participants) | 100
Number analyzed (Lesions) | 119
mm | 2.69 (0.43)

18. Secondary Outcome: In-segment Minimum Lumen Diameter (MLD)
Description: As measured by an independent angiographic core laboratory using quantitative coronary angiography (QCA); the minimum lumen diameter (MLD) measured at the in-segment region (in-segment includes the stented region and 5 mm edge regions).
  The MLD is the mean minimum lumen diameter (mm) from 2 orthogonal views.
Time Frame: Participants will be followed for the duration of hospital stay, an expected average of 1 day
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Lesions
Arm/Group | NG PROMUS Stent
Number analyzed (Participants) | 100
Number analyzed (Lesions) | 119
mm | 2.31 (0.46)

19. Secondary Outcome: Acute Gain
Description: Acute gain, as measured by angiographic core lab
Time Frame: Participants will be followed for the duration of hospital stay, an expected average of 1 day
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | NG PROMUS Stent
Number analyzed (Participants) | 100
mm | 1.84 (0.45)

20. Secondary Outcome: Vessel Area
Description: As measured by IVUS, the mean vessel area (mm2).
Time Frame: Participants will be followed for the duration of hospital stay, an expected average of 1 day
Measure: Mean (Standard Deviation); unit: mm^2
Units Other Than Participants: Lesions
Arm/Group | NG PROMUS Stent
Number analyzed (Participants) | 100
Number analyzed (Lesions) | 99
mm^2 | 15.1 (4.34)

21. Secondary Outcome: Stent Area
Description: As measured by IVUS, the area of the stent.
Time Frame: Participants will be followed for the duration of hospital stay, an expected average of 1 day
Measure: Mean (Standard Deviation); unit: mm^2
Units Other Than Participants: Lesions
Arm/Group | NG PROMUS Stent
Number analyzed (Participants) | 100
Number analyzed (Lesions) | 101
mm^2 | 7.83 (2.38)

22. Secondary Outcome: Lumen Area
Description: As measured by IVUS, the area of the lumen.
Time Frame: Participants will be followed for the duration of hospital stay, an expected average of 1 day
Measure: Mean (Standard Deviation); unit: mm^2
Units Other Than Participants: Lesions
Arm/Group | NG PROMUS Stent
Number analyzed (Participants) | 100
Number analyzed (Lesions) | 100
mm^2 | 7.76 (2.25)

23. Secondary Outcome: Vessel Volume
Description: As measured by IVUS, the volume of the vessel.
Time Frame: Participants will be followed for the duration of hospital stay, an expected average of 1 day
Measure: Mean (Standard Deviation); unit: mm^3
Units Other Than Participants: Lesions
Arm/Group | NG PROMUS Stent
Number analyzed (Participants) | 100
Number analyzed (Lesions) | 99
mm^3 | 354.34 (181.6)

24. Secondary Outcome: Stent Volume
Description: As measured by IVUS, the volume of the stent.
Time Frame: Participants will be followed for the duration of hospital stay, an expected average of 1 day
Measure: Mean (Standard Deviation); unit: mm^3
Units Other Than Participants: Lesions
Arm/Group | NG PROMUS Stent
Number analyzed (Participants) | 100
Number analyzed (Lesions) | 101
mm^3 | 185.3 (91.75)

25. Secondary Outcome: Lumen Volume
Description: As measured by IVUS, the volume of the lumen.
Time Frame: Participants will be followed for the duration of hospital stay, an expected average of 1 day
Measure: Mean (Standard Deviation); unit: mm^3
Units Other Than Participants: Lesions
Arm/Group | NG PROMUS Stent
Number analyzed (Participants) | 100
Number analyzed (Lesions) | 100
mm^3 | 182.6 (87.93)

26. Secondary Outcome: Incomplete Apposition
Description: Incomplete apposition rate, as measured by the IVUS core lab.
  Binary assessment of presence of one or more stent struts separated from the vessel wall as detected through intravascular ultrasound (IVUS).
Time Frame: Participants will be followed for the duration of hospital stay, an expected average of 1 day
Measure: Number; unit: percentage of lesions
Units Other Than Participants: Lesions
Arm/Group | NG PROMUS Stent
Number analyzed (Participants) | 100
Number analyzed (Lesions) | 101
percentage of lesions | 12.9

27. Secondary Outcome: Percent Net Volume Obstruction
Description: The percentage of volume obstruction, as measured by the IVUS core lab.
Time Frame: Participants will be followed for the duration of hospital stay, an expected average of 1 day
Measure: Mean (Standard Deviation); unit: % of volume
Units Other Than Participants: Lesions
Arm/Group | NG PROMUS Stent
Number analyzed (Participants) | 100
Number analyzed (Lesions) | 100
% of volume | 0 (.01)

28. Secondary Outcome: Longitudinal Stent Deformation
Description: Longitudinal stent deformation, evidenced by longitudinal compression or elongation, as the result of crossing a newly deployed stent with a second device, (such as a balloon catheter, stent system or IVUS catheter), causing the second device to become caught on the stent when the second device is advanced or retracted.
Time Frame: Participants will be followed for the duration of hospital stay, an expected average of 1 day
Measure: Number; unit: percentage of stents
Arm/Group | NG PROMUS Stent
Number analyzed (Participants) | 100
percentage of stents | 0

ADVERSE EVENTS:
Time Frame: Serious and non-serious adverse events were collected from the point of subject enrollment through study completion at 30 days.
Arm/Group | NG PROMUS Stent
Serious Adverse Events (participants affected / at risk) | 16/100
Other Adverse Events (participants affected / at risk) | 27/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NG PROMUS Stent (N=100)
Coronary artery dissection (Cardiac disorders) | 4 (4)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 1 (1)
Pericarditis (Cardiac disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 7 (7)
Pneumonia (Infections and infestations) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1)
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NG PROMUS Stent (N=100)
Myocardial infarction (Cardiac disorders) | 16 (16)
Coronary artery dissection (Cardiac disorders) | 5 (5)
Catheter site haematoma (General disorders) | 3 (3)
Presyncope (Nervous system disorders) | 2 (2)
Bradycardia (Cardiac disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Catheter site haemorrhage (General disorders) | 1 (1)
Procedural hypotension (Injury, poisoning and procedural complications) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1)
Blood urine present (Investigations) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Increased tendency to bruise (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution and Investigator shall have the right to publish the results, provided that before publishing, Institution and Investigator shall submit copies of any proposed publication or presentation to Sponsor for review at least sixty (60) days in advance of submission for publication or presentation to a publisher or other third party. Sponsor reserves the right to delete any confidential information or other proprietary information of Sponsor from the proposed publication or presentation.